CLINICAL TRIAL: NCT02131597
Title: Phase 2 Study of SGI-110 in Patients With Higher Risk MDS
Brief Title: Guadecitabine in Treating Patients With Higher-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0901; NCI-2014-02377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0901 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: High Risk Myelodysplastic Syndrome
MeSH Terms: interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (guadecitabine) (Experimental): Patients receive guadecitabine SC on days 1-5. Treatment repeats every 4-8 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 3 courses are taken off therapy after 6 courses. Patients may continue to receive treatment after 24 courses if the investigator determines it is in the patient's best interest.
  Interventions: Drug: Guadecitabine

INTERVENTIONS:
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110

SUMMARY:
This phase II trial studies how well guadecitabine works in treating patients with myelodysplastic syndromes that are at higher risk for becoming acute myeloid leukemia. Guadecitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the complete response (CR) rate with SGI-110 (guadecitabine) in patients with higher risk myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. Overall response rate, survival, transformation to acute myeloid leukemia (AML), transfusion independence.

II. Safety and toxicity.

OUTLINE:

Patients receive guadecitabine subcutaneously (SC) on days 1-5. Treatment repeats every 4-8 weeks for up to 24 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 3 courses are taken off therapy after 6 courses. Patients may continue to receive treatment after 24 courses if the investigator determines it is in the patient's best interest.

After completion of study treatment, patients are followed up at 30 days, and then every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with higher risk MDS (International Prognostic Scoring System [IPSS] int-2 or high; or >= 10% blasts as defined by World Health Organization [WHO])

  * No prior intensive chemotherapy or high-dose cytarabine (>= 1 g/m^2)
  * Prior biologic therapies (=< 1 cycle of prior decitabine or azacitidine), targeted therapies, or single agent chemotherapy is allowed
  * Off chemotherapy for 2 weeks prior to entering this study with no toxic effects of that therapy, unless there is evidence of rapidly progressive disease
  * Hydroxyurea is permitted for control of counts prior to treatment
  * Hematopoietic growth factors are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Serum creatinine =< 1.5 mg/dL
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST) or alanine transaminase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Provide signed written informed consent
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Female patients of childbearing potential must have a negative pregnancy test within 2 weeks prior to entering this study
* Women who are able to become pregnant and men who can father a child must use birth control while on study and for at least 8 weeks after your last dose of study drug(s); acceptable birth control includes a condom or a diaphragm with spermicidal jelly; and birth control methods that are taken by mouth, injected, or implanted; if you are already using birth control, you must check with the study staff to make sure that it is considered one of the acceptable forms to use in this study

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks prior to entering this study with the exception of hydroxyurea; the patient must have recovered from all acute toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Any concurrent malignancy

  * Exceptions

    * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed
    * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11-10 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Urrutia S, Bose P, Alvarado Y, Borthakur G, Ravandi F, Daver N, Pemmaraju N, Jabbour E, Takahashi K, Kadia T, DiNardo C, Kornblau S, Kanagal-Shamanna R, Huang X, Bodden K, Kantarjian H, Garcia-Manero G. Prospective performance of the IWG-2023 criteria and IPSS-M in a phase 2 trial of guadecitabine for higher-risk MDS or CMML. Blood Neoplasia. 2024 Mar 29;1(2):100008. doi: 10.1016/j.bneo.2024.100008. eCollection 2024 Jun. PMID 40454402
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Guadecitabine)
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Guadecitabine)
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 66
Age, Continuous [Median (Full Range); unit: years] | 69 [22 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 87
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response (CR)
Description: Complete Response is Normalization of the peripheral blood and bone marrow with </= 5% bone marrow blasts, a peripheral blood granulocyte count >/= 1.0 x 10^9/L, and a platelet count >/= 100 x 10^9/L. Hemoglobin >/= 11 g/dL at any point while on treatment after the first cycle of therapy.
Time Frame: At cycle 3 and cycle 6, cycles are up every 4 to 8 weeks. Up to 9 years, 8 months and 15 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Guadecitabine)
Number analyzed (Participants) | 100
Participants | 25

2. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 9 years, 8 months and 15 days
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Guadecitabine)
Number analyzed (Participants) | 100
Months | 16.9 [1.0 to 59.3]

3. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Transformation
Time Frame: Up to 9 years, 8 months and 15 days
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Guadecitabine)
Number analyzed (Participants) | 100
Months | 27.3 [0.96 to 69.9]

ADVERSE EVENTS:
Time Frame: Up to 9 years, 8 months and 15 days
Arm/Group | Treatment (Guadecitabine)
All-Cause Mortality (participants affected / at risk) | 14/100
Serious Adverse Events (participants affected / at risk) | 76/100
Other Adverse Events (participants affected / at risk) | 93/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Guadecitabine) (N=100)
Abdominal pain (General disorders) | 3 (3)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1)
Acute coronary syndrome (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (3)
Bacteremia (Infections and infestations) | 10 (12)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiopulomary Arrest (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 6 (6)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Clostridium difficile (Infections and infestations) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Device-related infection (Infections and infestations) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (30)
Flu-like symptoms (General disorders) | 1 (1)
Fungal Pneumonia (Infections and infestations) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Heart Failure (Cardiac disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hepatic infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 5 (6)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Non-cardiac chest pain (Cardiac disorders) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Penumonia (Infections and infestations) | 10 (11)
Peripheral vascular occlusive disease (Vascular disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Pneumonia (Infections and infestations) | 9 (12)
Retinal vascular disorder (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 6 (8)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Soft tissue infection (Infections and infestations) | 3 (3)
Stroke (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (6)
Thromboembolic Event (Vascular disorders) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 7 (7)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
GI perforation (Gastrointestinal disorders) | 1 (1)
muscle abscess (Infections and infestations) | 1 (1)
Fungal sinusitis (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Guadecitabine) (N=100)
Upper respiratory infection (Infections and infestations) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 5 (6)
Skin infection (Infections and infestations) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Fever (General disorders) | 7 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (7)
Hypotension (Vascular disorders) | 7 (7)
Pain (General disorders) | 5 (8)
Urinary tract infection (Infections and infestations) | 8 (9)
Edema limbs (General disorders) | 5 (10)
Dizziness (Nervous system disorders) | 7 (11)
Neutrophil count decreased (Investigations) | 9 (11)
Headache (Nervous system disorders) | 8 (12)
Vomiting (Gastrointestinal disorders) | 11 (13)
Diarrhea (Gastrointestinal disorders) | 15 (15)
White blood cell decreased (Investigations) | 9 (16)
Infections and infestations (Infections and infestations) | 15 (18)
Constipation (Gastrointestinal disorders) | 17 (23)
Mucositis oral (Gastrointestinal disorders) | 17 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (30)
Injection site reaction (General disorders) | 19 (30)
Platelet count decreased (Infections and infestations) | 14 (30)
Lung infection (Infections and infestations) | 28 (34)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (35)
Nausea (Gastrointestinal disorders) | 30 (40)
Fatigue (General disorders) | 52 (105)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT02131597/Prot_SAP_000.pdf